CLINICAL TRIAL: NCT04465357
Title: A Multicenter, Open Label Study Assessing the Efficacy of Erenumab on Functional Impact of Migraine
Brief Title: Efficacy of Erenumab on Functional Impact of Migraine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merle Diamond (Other)
Collaborators: Clinvest Research, LLC (Industry); Smith, Timothy R., M.D. (Individual)
Responsible Party: Sponsor-Investigator, Merle Diamond, President, Managing Director, Diamond Headache Clinic
Organization: Diamond Headache Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-001AM
Record Dates: First submitted 2020-07-07; First posted 2020-07-10 (Actual); Results first posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-09

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — erenumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Erenumab-Aooe 140 MG/ML [Aimovig] (Experimental): Participants received 140 mg/mL administered subcutaneously once every 4 weeks in the abdomen, thigh, or upper arm for three months (12 weeks).
  Interventions: Drug: Erenumab-Aooe 140 MG/ML [Aimovig]

INTERVENTIONS:
Drug: Erenumab-Aooe 140 MG/ML [Aimovig] — 140 mg/mL administered subcutaneously
  Other Names: Erenumab; Aimovig

SUMMARY:
The purpose of this study is to assess the efficacy of erenumab on functional impact due to Migraine in adults.

DETAILED DESCRIPTION:
This is a single group, multicenter, open-label study with a study population of patients who meet International Classification of Headache Disorders 3rd edition (ICHD-III) criteria for migraine with or without aura and have 4 to 20 migraine days per month. This is a single-group supportive care study with one arm and no masking. A maximum of 54 participants will be enrolled to study intervention. All participants in this single-group study will complete a 4-week run-in period. After the run-in period, eligible participants will be enrolled to study intervention and enter a 12-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

1. willing to participate and sign informed consent;
2. ability to understand informed consent and study procedures, including able to use the electronic Daily Headache Diary;
3. in good general health based on investigator's judgment;
4. must be between 18 to 65 years of age, inclusive, at time of Visit 2;
5. have migraine with or without aura meeting the diagnostic criteria listed in the International Classification of Headache Disorders 3rd edition (ICHD-III; Appendix 5);
6. verification of headache frequency through prospectively collected baseline information during the 28-day screening/baseline phase reporting 4-20 migraine days and no more than 20 total headache days;
7. onset of migraine before age 50;
8. able to differentiate migraine from other primary headache types allowed in the study (e.g., tension-type headache);
9. stable history of migraine at least 3 months prior to screening with headache free periods;
10. not currently taking a migraine preventive OR has been taking a stable dose of a preventive for at least 90 days prior to screening and agrees to not start, stop, or change medication and/or dosage during the study period;

    **participants on migraine preventive should have stable headache pattern
11. must have a score of ≥ 3 on the Migraine Functional Impact Questionnaire (MFIQ) overall impact on usual activities item at screening;
12. women may be included only if they have a negative pregnancy test at screening and baseline, are sterile, or postmenopausal. Women of childbearing potential (WOCBP) whose male partners are potentially fertile (i.e., no vasectomy) must use highly effective birth control methods for the duration of the study (i.e., starting at screening). Definitions of WOCBP, sterile and postmenopausal women, male contraception, and highly effective and acceptable birth control methods are to be determined based on investigator's judgment;
13. demonstrated compliance with the electronic Daily Headache Diary during the 28-day screening/baseline phase as defined by entry of headache data on a minimum of 23 days;
14. is willing to wear activity/sleep tracker throughout the duration of the trial;
15. has a smartphone and willing to install activity tracker app on phone.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. unable to understand the study requirements, the informed consent, or complete headache records as required per protocol;
2. pregnant, actively trying to become pregnant, or breast-feeding;
3. history of substance abuse and/or dependence, in the opinion of the Investigator;
4. history of impaired renal function that, in the investigator's opinion, contraindicates participation in this study;
5. suffers from a serious illness, or an unstable medical condition, one that could require hospitalization, or could increase the risk of adverse events;
6. a psychiatric condition, in the opinion of the investigator, that may affect the interpretation of efficacy and safety data or contraindicates the participant's participation in the study;
7. received nerve blocks or trigger point injections in the previous 8 weeks or plans to receive them during the study;
8. prior exposure in the last 6 months to biologics or drugs specifically targeting the calcitonin gene-related peptide (CGRP) pathway;
9. has failed more than 3 classes of medications for the prevention of migraine, or >6 migraine preventative medications of any type due to lack of efficacy;
10. received any investigational agents within 30 days prior to Visit 1 (6 months for any investigational biological products unless previous study blind has been broken and subject was known to have received placebo);
11. plans to participate in another clinical study at any time during this study;
12. history of medication overuse of opioids or butalbital, as defined by opioid or butalbital use ≥10 days/month in previous 12 months or during run-in period; Medication Overuse Headache (MOH) with other medication types will be allowed but must be documented;
13. unstable medication use for migraine prevention (changes in the last 3 months);
14. clinically relevant lab results at screening as determine by the investigator;
15. clinically relevant or significant ECG abnormalities as determine by the investigator, including ECG with QT interval corrected for heart rate (QTc) using Fridericia's correction formula (QTcF) > 500 msec;
16. history of any of the following cardiovascular conditions:

    1. Moderate to severe congestive heart failure (New York Heart Association class III or IV);
    2. Recent (within past 12 months) cerebrovascular accident, myocardial infarction, coronary stenting;
    3. Uncontrolled hypertension as defined by a confirmed systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg.
17. active HIV or Hepatitis C infection;
18. allergy to latex;
19. score of > 0 on question 9 on Patient Health Questionnaire (PHQ-9) at any visit;
20. have any other condition, that in the judgment of the investigator, would make the participant unsuitable for inclusion, or would interfere with the participant participating in or completing the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merle Diamond, MD, Principal Investigator — Diamond Headache Clinic
Locations (3):
- United States (3):
  - Diamond Headache Clinic, Chicago, Illinois
  - StudyMetrix, City of Saint Peters, Missouri
  - Clinvest Research, Springfield, Missouri

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erenumab-Aooe 140 MG/ML [Aimovig]
Started | 55
Completed | 42
Not Completed | 13
Not completed — Adverse Event | 2
Not completed — Lack of Efficacy | 1
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 6
Not completed — Protocol specified withdrawal criterion met | 2

BASELINE CHARACTERISTICS:
Arm/Group | Erenumab-Aooe 140 MG/ML [Aimovig]
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.35 (11.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 52
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 52
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 55
MFIQ Global Item [Mean (Standard Deviation); unit: units on a scale] — The MFIQ is a 26-item self-report questionnaire. A single global item assess overall difficulty doing everyday activities. Final transformed scores range from 0-100, with higher scores indicating more impact on the participant.
  units on a scale | 43.64 (23.18)
Monthly Migraine Days [Mean (Standard Deviation); unit: Days per month] — Number of days per month with Migraine (with or without Aura) as defined by ICHD-3 criteria.
  Days per month | 10.01 (3.90)

OUTCOME MEASURES:

1. Primary Outcome: Migraine Functional Impact Questionnaire (MFIQ) - "Overall Impact on Usual Activities" Scores at Baseline and at End of Treatment (Treatment Month 3).
Description: The Migraine Functional Impact Questionnaire (MFIQ) is a 26-item self-report questionnaire. It is designed to measure the impact of migraine on physical, social, and emotional functioning over 5 domains: Physical Function (PF), Usual Activities (UA), Overall impact on Usual Activities, Social Function (SF), and Emotional Function (EF). Final transformed scores range from 0-100, with higher scores indicating more impact on the participant. For this endpoint we will be measuring changes in participant's response on the single MFIQ Global Item Overall Impact on Usual Activities (item # 16). The item's transformed score can range from 0-100, with higher scores indicating more impact on the participant.
Time Frame: Baseline and Treatment Month 3
Population: Full analysis population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Erenumab-Aooe 140 MG/ML [Aimovig]
Number analyzed (Participants) | 55
score on a scale
  Baseline | 43.64 (23.18)
  Treatment Month 3 | 21.82 (20.44)

2. Secondary Outcome: Migraine Functional Impact Questionnaire (MFIQ) - "Impact on Physical Function" Domain Scores at Baseline and at the End of Treatment (Treatment Month 3).
Description: The Migraine Functional Impact Questionnaire (MFIQ) is a 26-item self-report questionnaire. It is designed to measure the impact of migraine on physical, social, and emotional functioning over 5 domains: Physical Function (PF), Usual Activities (UA), Overall impact on Usual Activities, Social Function (SF), and Emotional Function (EF). Final transformed scores range from 0-100, with higher scores indicating more impact on the participant. For this endpoint we will be measuring changes in participant's response on the MFIQ domain, Physical Function. The domain's transformed score can range from 0-100, with higher scores indicating more impact on the participant.
Time Frame: Baseline and Treatment Month 3
Population: Full analysis population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Erenumab-Aooe 140 MG/ML [Aimovig]
Number analyzed (Participants) | 55
score on a scale
  Baseline | 48.82 (17.56)
  Treatment Month 3 | 25.84 (21.41)

3. Secondary Outcome: Migraine Functional Impact Questionnaire (MFIQ) - "Impact on Usual Activities" Scores at Baseline and at the End of Treatment (Treatment Month 3).
Description: The Migraine Functional Impact Questionnaire (MFIQ) is a 26-item self-report questionnaire. It is designed to measure the impact of migraine on physical, social, and emotional functioning over 5 domains: Physical Function (PF), Usual Activities (UA), Overall impact on Usual Activities, Social Function (SF), and Emotional Function (EF). Final transformed scores range from 0-100, with higher scores indicating more impact on the participant. For this endpoint we will be measuring changes in participant's response on the MFIQ domain, Usual Activities. The domain's transformed score can range from 0-100, with higher scores indicating more impact on the participant.
Time Frame: Baseline and Treatment Month 3
Population: Full analysis population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Erenumab-Aooe 140 MG/ML [Aimovig]
Number analyzed (Participants) | 55
score on a scale
  Baseline | 39.16 (21.36)
  Treatment Month 3 | 17.81 (18.36)

4. Secondary Outcome: Migraine Functional Impact Questionnaire (MFIQ) - "Impact on Emotional Function" Scores at Baseline and at the End of Treatment (Treatment Month 3).
Description: The Migraine Functional Impact Questionnaire (MFIQ) is a 26-item self-report questionnaire. It is designed to measure the impact of migraine on physical, social, and emotional functioning over 5 domains: Physical Function (PF), Usual Activities (UA), Overall impact on Usual Activities, Social Function (SF), and Emotional Function (EF). Final transformed scores range from 0-100, with higher scores indicating more impact on the participant. For this endpoint we will be measuring changes in participant's response on the MFIQ domain, Emotional Function. The domain's transformed score can range from 0-100, with higher scores indicating more impact on the participant.
Time Frame: Baseline and Treatment Month 3
Population: Full analysis population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Erenumab-Aooe 140 MG/ML [Aimovig]
Number analyzed (Participants) | 55
score on a scale
  Baseline | 43.00 (27.67)
  Treatment Month 3 | 19.64 (22.13)

5. Secondary Outcome: Migraine Functional Impact Questionnaire (MFIQ) - "Impact on Social Function" Scores at Baseline and at the End of Treatment (Treatment Month 3).
Description: The Migraine Functional Impact Questionnaire (MFIQ) is a 26-item self-report questionnaire. It is designed to measure the impact of migraine on physical, social, and emotional functioning over 5 domains: Physical Function (PF), Usual Activities (UA), Overall impact on Usual Activities, Social Function (SF), and Emotional Function (EF). Final transformed scores range from 0-100, with higher scores indicating more impact on the participant. For this endpoint we will be measuring changes in participant's response on the MFIQ domain, Social Function. The domain's transformed score can range from 0-100, with higher scores indicating more impact on the participant.
Time Frame: Baseline and Treatment Month 3
Population: Full analysis population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Erenumab-Aooe 140 MG/ML [Aimovig]
Number analyzed (Participants) | 55
score on a scale
  Baseline | 40.36 (21.49)
  Treatment Month 3 | 17.86 (20.52)

6. Secondary Outcome: Migraine Functional Impact Questionnaire (MFIQ) - "Overall Impact on Usual Activities" Scores at Baseline and at Treatment Months 1, 2, and 3.
Description: as for outcome 1
Time Frame: Baseline and Treatment Months 1, 2, and 3
Population: Full analysis population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Erenumab-Aooe 140 MG/ML [Aimovig]
Number analyzed (Participants) | 55
score on a scale
  Baseline | 43.64 (23.18)
  Treatment Month 1 | 23.18 (21.44)
  Treatment Month 2 | 23.18 (23.50)
  Treatment Month 3 | 21.82 (20.44)

7. Secondary Outcome: Migraine Functional Impact Questionnaire (MFIQ) - "Impact on Physical Function" Scores at Baseline and at Treatment Months 1, 2, and 3.
Description: The Migraine Functional Impact Questionnaire (MFIQ) is a 26-item self-report questionnaire. It is designed to measure the impact of migraine on physical, social, and emotional functioning over 5 domains: Physical Function (PF), Usual Activities (UA), Overall impact on Usual Activities, Social Function (SF), and Emotional Function (EF). Final transformed scores range from 0-100, with higher scores indicating more impact on the participant. For this endpoint we will be measuring changes in participant's response on the MFIQ domain, Physical Function The domain's transformed score can range from 0-100, with higher scores indicating more impact on the participant.
Time Frame: Baseline and Treatment Months 1, 2, and 3
Population: Full Analysis population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Erenumab-Aooe 140 MG/ML [Aimovig]
Number analyzed (Participants) | 55
score on a scale
  Baseline | 48.82 (17.56)
  Treatment Month 1 | 29.34 (23.10)
  Treatment Month 2 | 28.91 (23.74)
  Treatment Month 3 | 25.84 (21.41)

8. Secondary Outcome: Migraine Functional Impact Questionnaire (MFIQ) - "Impact on Usual Activities" Scores at Baseline and at Treatment Months 1, 2, and 3.
Description: as for outcome 3
Time Frame: Baseline and Treatment Months 1, 2, and 3
Population: Full analysis population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Erenumab-Aooe 140 MG/ML [Aimovig]
Number analyzed (Participants) | 55
score on a scale
  Baseline | 39.6 (21.36)
  Treatment Month 1 | 21.18 (20.50)
  Treatment Month 2 | 20.02 (21.73)
  Treatment Month 3 | 17.81 (18.36)

9. Secondary Outcome: Migraine Functional Impact Questionnaire (MFIQ) - "Impact on Emotional Function" Scores at Baseline and at Treatment Months 1, 2, and 3.
Description: as for outcome 4
Time Frame: Baseline and Treatment Months 1, 2, and 3
Population: Full Analysis population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Erenumab-Aooe 140 MG/ML [Aimovig]
Number analyzed (Participants) | 55
score on a scale
  Baseline | 43.00 (27.67)
  Treatment Month 1 | 22.00 (24.39)
  Treatment Month 2 | 21.55 (25.42)
  Treatment Month 3 | 19.64 (22.13)

10. Secondary Outcome: Migraine Functional Impact Questionnaire (MFIQ) - "Impact on Social Function" Scores at Baseline and at Treatment Months 1, 2, and 3.
Description: as for outcome 5
Time Frame: Baseline and Treatment Months 1, 2, and 3
Population: Full Analysis Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Erenumab-Aooe 140 MG/ML [Aimovig]
Number analyzed (Participants) | 55
score on a scale
  Baseline | 40.36 (21.49)
  Treatment Month 1 | 18.55 (20.96)
  Treatment Month 2 | 18.98 (22.75)
  Treatment Month 3 | 17.86 (20.52)

11. Secondary Outcome: Migraine Interictal Burden Scale (MIBS-4) Scores at Baseline and at Treatment Months 1, 2, and 3.
Description: The Migraine Interictal Burden Scale (MIBS-4) is a 4-item, self-administered questionnaire which measures interictal migraine-related burden in 4 domains: impairment in work or school, impairment in family and social life, difficulty making plans or commitments, and emotional/affective and cognitive distress. Possible scores range from 0 (No interictal burden) to 12 (Severe interictal burden). Higher scores indicate worse interictal burden.
Time Frame: Baseline and Treatment Months 1, 2, and 3
Population: Full Analysis Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Erenumab-Aooe 140 MG/ML [Aimovig]
Number analyzed (Participants) | 55
score on a scale
  Baseline | 5.11 (3.23)
  Treatment Month 1 | 3.44 (3.09)
  Treatment Month 2 | 3.31 (3.05)
  Treatment Month 3 | 3.00 (3.03)

12. Secondary Outcome: Number of Migraine Days at Baseline and at Treatment Months 1, 2, and 3.
Description: Comparison of the mean change from baseline in the frequency of migraine headache days per 28-day period ending with the cessation of treatment month 3. A migraine headache day will be defined as a calendar day (00:00 to 23:59) with 4 or more hours of migraine headache, fulfilling International Classification of Headache Disorders-3 criteria, and/or any headache of any duration with the use of migraine-specific acute medications(s) (i.e. ergot alkaloids, ergot combinations, opioids, triptans, combination analgesics [simple analgesics combined with opioids or barbiturate with or without caffeine]).
Time Frame: Baseline and Treatment Months 1, 2, and 3
Population: Full Analysis Population
Measure: Mean (Standard Deviation); unit: days per month
Arm/Group | Erenumab-Aooe 140 MG/ML [Aimovig]
Number analyzed (Participants) | 55
days per month
  Baseline | 10.06 (3.90)
  Treatment Month 1 | 7.82 (5.13)
  Treatment Month 2 | 6.96 (4.60)
  Treatment Month 3 | 6.33 (4.64)

13. Secondary Outcome: Work Productivity and Activity Impairment- Migraine (WPAI-M): Absenteeism Domain Scores at Baseline and at Treatment Months 1, 2, and 3.
Description: The Work Productivity and Activity Impairment- Migraine (WPAI-M) is a 6-item self-administered questionnaire that measures work productivity and the amount of time missed from work due to migraine. Domain scores are expressed as a percentage, with a range of scores form 0-100%, with higher scores indicating greater impairment and less productivity.
Time Frame: Baseline and Treatment Months 1, 2, and 3
Population: Full Analysis population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Erenumab-Aooe 140 MG/ML [Aimovig]
Number analyzed (Participants) | 55
score on a scale
  Baseline | 9.11 (13.02)
  Treatment Month 1 | 3.50 (7.10)
  Treatment Month 2 | 4.43 (9.80)
  Treatment Month 3 | 3.09 (6.76)

14. Secondary Outcome: Work Productivity and Activity Impairment- Migraine (WPAI-M): Activity Impairment Domain Scores at Baseline and at Treatment Months 1, 2, and 3.
Description: as for outcome 13
Time Frame: Baseline and Treatment Months 1, 2, and 3
Population: Full Analysis population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Erenumab-Aooe 140 MG/ML [Aimovig]
Number analyzed (Participants) | 55
score on a scale
  Baseline | 52.18 (25.94)
  Treatment Month 1 | 31.82 (27.83)
  Treatment Month 2 | 25.82 (26.30)
  Treatment Month 3 | 26.00 (25.86)

15. Secondary Outcome: Work Productivity and Activity Impairment- Migraine (WPAI-M): Work Productivity Loss Domain Scores at Baseline and at Treatment Months 1, 2, and 3.
Description: as for outcome 13
Time Frame: Baseline and Treatment Months 1, 2, and 3
Population: Full Analysis population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Erenumab-Aooe 140 MG/ML [Aimovig]
Number analyzed (Participants) | 55
score on a scale
  Baseline | 48.12 (25.04)
  Treatment Month 1 | 30.09 (24.55)
  Treatment Month 2 | 27.90 (24.83)
  Treatment Month 3 | 22.79 (24.85)

16. Secondary Outcome: Work Productivity and Activity Impairment- Migraine (WPAI-M): Presenteeism Domain Scores at Baseline and at Treatment Months 1, 2, and 3.
Description: as for outcome 13
Time Frame: Baseline and Treatment Months 1, 2, and 3
Population: Full Analysis population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Erenumab-Aooe 140 MG/ML [Aimovig]
Number analyzed (Participants) | 55
score on a scale
  Baseline | 48.07 (21.82)
  Treatment Month 1 | 30.32 (22.73)
  Treatment Month 2 | 26.77 (22.42)
  Treatment Month 3 | 23.23 (23.58)

17. Secondary Outcome: Neuro-QoL Sleep Disturbance Short Form (SDSF) Scores at Baseline and at Treatment Months 1, 2, and 3.
Description: The Neuro-QoL Sleep Disturbance Short Form (SDSF) is an 8-item, self-administered questionnaire which measures quality of sleep including difficulties and perception of sleep satisfaction. Possible transformed t-scores ranging from 32 to 84.20, with higher scores indicating worse sleep habits.
Time Frame: Baseline and Treatment Months 1, 2, and 3
Population: Full Analysis population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Erenumab-Aooe 140 MG/ML [Aimovig]
Number analyzed (Participants) | 55
score on a scale
  Baseline | 56.58 (7.04)
  Treatment Month 1 | 52.50 (8.14)
  Treatment Month 2 | 52.89 (7.72)
  Treatment Month 3 | 50.93 (9.40)

18. Secondary Outcome: General Self-Efficacy Severity Scale (GSESS) Scores at Baseline and at Treatment Months 1, 2, and 3.
Description: The General Self-Efficacy Severity Scale (GSESS) is a 4 item, self-administered questionnaire where the participant is asked to rate their confidence in managing situations, problems, and events. Final scores range from 18.60 to 64.70 and are represented by the T-score, a standardized score with a mean of 50 and a standard deviation (SD) of 10. Higher scores indicate the participant has more self-efficacy managing difficult situations.
Time Frame: Baseline and Treatment Months 1, 2, and 3
Population: Full Analysis population
Measure: Mean (Standard Deviation); unit: T-Scores
Arm/Group | Erenumab-Aooe 140 MG/ML [Aimovig]
Number analyzed (Participants) | 55
T-Scores
  Baseline | 50.20 (8.83)
  Treatment Month 1 | 53.42 (8.13)
  Treatment Month 2 | 52.95 (8.75)
  Treatment Month 3 | 54.87 (8.42)

19. Secondary Outcome: Brief Measure of Worry Severity (BMWS) Scores at Baseline and at Treatment Months 1, 2, and 3
Description: The Brief Measure of Worry Severity (BMWS) is a 8-item, self-administered questionnaire that measures various components of dysfunctional worry. Score range from 0-24 with higher scores indicating more worry within the participant.
Time Frame: Baseline and Treatment Months 1, 2, and 3
Population: Full Analysis population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Erenumab-Aooe 140 MG/ML [Aimovig]
Number analyzed (Participants) | 55
score on a scale
  Baseline | 7.42 (5.87)
  Treatment Month 1 | 5.84 (5.17)
  Treatment Month 2 | 5.75 (5.19)
  Treatment Month 3 | 5.16 (5.09)

ADVERSE EVENTS:
Time Frame: 12 weeks (from Visit 2 [enrollment visit] to Visit 5 [end of study])
Arm/Group | Erenumab-Aooe 140 MG/ML [Aimovig]
All-Cause Mortality (participants affected / at risk) | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55
Other Adverse Events (participants affected / at risk) | 3/55
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erenumab-Aooe 140 MG/ML [Aimovig] (N=55)
Constipation (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Per contractual agreement PIs agree to submit drafts of all publications to sponsor and funding sponsor between a period of 5 and 45 days depending on publication type (e.g. manuscript, poster, etc.).

DOCUMENTS (2):
  • Study Protocol (2020-09-16): https://cdn.clinicaltrials.gov/large-docs/57/NCT04465357/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-23): https://cdn.clinicaltrials.gov/large-docs/57/NCT04465357/SAP_001.pdf